CLINICAL TRIAL: NCT00387985
Title: An Open-label, Single-dose, Randomized, 2-period Crossover, Bioequivalence Study Between the Current Formulation and the New Formulation of MOA-728 Administered Subcutaneously in Healthy Subjects
Brief Title: Bioequivalence Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3200K1-103
Record Dates: First submitted 2006-10-11; First posted 2006-10-13 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Healthy

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
Primary: To determine the bioequivalence between the new formulation and the current formulation of the investigational drug, MOA-728.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Willingboro, New Jersey, United States